CLINICAL TRIAL: NCT01356303
Title: A Phase II Study of Docetaxel Combined With Cisplatin as the First Line Chemotherapy in Patients With Metastatic Non-small Cell Lung Cancer
Brief Title: Docetaxel Combined With Cisplatin as First Line in Patients With Metastatic Non-small Cell Lung Cancer
Acronym: TAXIS01
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty in enrolling patients
Sponsor: National Guard Health Affairs (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC08/068
Record Dates: First submitted 2011-03-19; First posted 2011-05-19 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Non-small Cell Lung Cancer Metastatic
Keywords: Lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cisplatin, Docetaxel (Experimental): Each cycle of chemotherapy administration will be started with docetaxel at dose of 75 mg/m2 in 250 ml of D5W or NS administered as a 1-hour intravenous infusion, followed by cisplatin at dose of 75 mg/m2administered as a 2-hour intravenous infusion every 3 weeks per cycle for 4-6 cycles
  Interventions: Drug: cisplatin, docetaxel

INTERVENTIONS:
Drug: cisplatin, docetaxel — All patients met the eligibility criteria will undergo treatment with chemotherapy.
  Each cycle of chemotherapy administration will be started with docetaxel at dose of 75 mg/m2 in 250 ml of Dextrose 5% in Water or Normal Saline administered as a 1-hour intravenous infusion followed by cisplatin at dose of 75 mg/m2 administered as a 2-hour intravenous infusion every 3 weeks per cycle for totally 4-6 cycles.

SUMMARY:
This is a phase II, open-label clinical study prospectively enrolling 40 metastatic patients with non small cell lung cancer. The study will enroll patients at King Abdulaziz Medical City, Riyadh.

Sub-sites will be open for patient accrual in selected centers in the Kingdom.

DETAILED DESCRIPTION:
The cisplatin/docetaxel is established standard in the first line management of metastatic non small cell lung cancer in the United States, Europe and Asia. However, the safety and efficacy of this regimen was not studied systematically in Middle Eastern population. The aim of this study is to study the efficacy and safety of this regimen in our patient population

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven non-small cell lung carcinoma
* Stage IV metastatic non-small cell lung carcinoma or stage III with malignant pleural effusion.
* Patient should not be eligible for customization chemotherapy (if available at participating institutions).
* Having at least one measurable lesion
* Patient has life expectancy of 12 weeks or greater.
* Age > 18 years.
* No prior systemic treatment for metastatic lung cancer. Adjuvant treatment given more than 1 year ago is acceptable.
* WHO performance status 0-2 (See Appendix III )
* Adequate organ function:

  * Hematology: Neutrophils > 2 x 10 9 /L, platelets > 100 x 10 9 /L
  * Hepatic function: Total bilirubin < 1.25 times the upper normal limits, ASAT (SGOT) < 2 times the upper normal limits
  * Renal function: Creatinine < 1.5 mg/dL; if value is higher than upper normal limit but less than 2 mg/dL, the creatinine clearance should be > 60min/ml.
* Able to comply with scheduled follow-up and with management of toxicity
* Signed informed consent from patient or legal representative
* Negative urine pregnancy test (if indicated)

Exclusion Criteria:

* Pregnant or lactating women or women of childbearing potential using inadequate contraception.
* Uncontrolled brain metastatic disease. (CNS disease that is stable > 4 weeks after radiotherapy in lieu of steroids reduction is eligible).
* Symptomatic peripheral neuropathy > grade 1 according to the NCI Common Toxicity Criteria Version 3
* Other serious illness or medical condition:

  * Unstable cardiac disease requiring treatment
  * History of significant neurologic or psychiatric disorders including psychotic disorders, dementia or seizures
  * Active uncontrolled infection
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational drug within 30 days prior to study screening
* Concurrent treatment with any other anti-cancer therapy
* Contraindication of steroid drug administration
* Past (up to 5 years) or concurrent history of other neoplasm except curatively treated non- melanoma skin cancer or in situ carcinoma of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-03; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 3 years
  Efficacy will be measured by calculating the following:
  * Response rate using Response Evaluation Criteria for Solid Tumor criteria
  * Time to Disease progression or Death
  * Overall Survival

SECONDARY OUTCOMES:
Progression free survival, safety | 3 years
  * To determine progression free survival, median survival and 1 year survival of the studied population.
  * To evaluate the Number of participants with Adverse Events and Serious Adverse Events.Safety will include 4 parameters to be collected for all patients who receive the study regimen which are:
    * Adverse Events
    * Laboratory Assessments
    * Vital Signs
    * Physical Examinations

CONTACTS AND LOCATIONS:
Overall Officials: Abdulrahman Jazieh, MD/MPH, Principal Investigator — King Abdul Aziz Medical City for National Guard
Locations (1):
- King Abdul Aziz Medical City for National Guard Health Affairs, Riyadh, Saudi Arabia